CLINICAL TRIAL: NCT01147341
Title: Can TNF-Alpha Incomplete Secondary Responders Attain a Safe and Efficacious Response By Switching to Certolizumab Pegol (Cimzia)? A Phase IV, Randomized, Multi-Center, Double-Blind, Twelve-Week Study Followed by a 12-Week Open-Label Phase
Brief Title: Can TNF-Alpha Incomplete Secondary Responders Attain a Safe and Efficacious Response Switching to Cimzia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Schiff, MD (Individual)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Michael Schiff, MD, MD, Schiff, Michael, M.D.
Organization: Schiff, Michael, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CERT-001
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; anti-TNF therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Placebo (0.9% sodium chloride) given as 2 subcutaneous (sc) injections at weeks 0, 2, and 4, followed y 1 sc injection given an weeks 6, 8, and 10. At week 12 subjects entered the open label phase. Subjects received 400 mg of Cimzia (CZP) given as two 200 mg subcutaneous (sc) injections at weeks 12,14 and 16, followed by 1 sc injection at weeks 18, 20, and 22.
  Interventions: Drug: Placebo
- active treatment with Cimzia (Active Comparator): 400 mg of Cimzia (CZP) given as two 200 mg subcutaneous (sc) injections at weeks 0, 2, and 4, followed by 1 sc injection at weeks 6, 8, and 10. At week 12 subjects entered the open label phase. Subjects received 400 mg of Cimzia (CZP) given as two 200 mg subcutaneous (sc) injections at weeks 12,14 and 16, followed by 1 sc injection at weeks 18, 20, and 22.
  Interventions: Drug: Cimzia

INTERVENTIONS:
Drug: Cimzia — prefilled 200mg Cimzia syringe SC q 2 weeks
  Other Names: 1 ml liquid product containing 200mg of Certolizumab Pegol
  Arms: active treatment with Cimzia
Drug: Placebo — prefilled saline syringe
  Other Names: 1 ml Sodium Cloride 0.9%
  Arms: placebo

SUMMARY:
Purpose of the study is to determine if Cimzia is safe and effective in subjects who have received previous treatment with a TNF-alpha inhibitor other than Cimzia.

DETAILED DESCRIPTION:
This is a Phase IV, randomized, multi-center, double-blind, parallel-group 12-week study of Cimzia with concomitant methotrexate (MTX) or other DMARD compared to MTX or other DMARD alone in patients with an inadequate secondary therapeutic response to a TNF-alpha inhibitor as defined above and active rheumatoid arthritis (RA) followed by a 12-week open-label phase with concomitant MTX or other DMARD and Cimzia.

Subjects must washout from the previous TNF inhibitor for at least 4 weeks prior to the baseline visit. Subjects unable to tolerate MTX must have been on a stable dose of another non-biologic DMARD for at least 3 months. Subjects' diagnosis of RA must be based on the 1987 Revised American Rheumatism Association Criteria for the Classification of Rheumatoid Arthritis.

Subjects will be screened for eligibility and, up to 28 days later, at the baseline visit, randomized to one of two treatment groups (2:1): Cimzia or placebo (in addition to concomitant MTX or other DMARD). All subjects will continue MTX/other DMARD at the same dose utilized prior to study entry.

After the Week 12 study visit, all subjects will have the opportunity to continue in the study on open-label Cimzia treatment (using an induction regimen for all subjects, regardless of their treatment in the blinded phase).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of RA at least 6 months
* Have received treatment with a TNF-alpha inhibitor
* Be receiving Methotrexate (with folic acid)at a dose of at least 10mg/week or another non-biologic DMARD if Methotrexate intolerant *Have at least 6 tender joint and 6 swollen joints*
* Have an CRP greater than or equal to ULN
* Availability of a chest x-ray that shows no evidence of active TB or infection

Exclusion Criteria:

* Prior exposure to Cimzia
* Prior treatment with B-cell depleting therapy
* No significant response to previous TNF inhibitor
* Congestive heart failure
* Clinically abnormal laboratory tests
* History of cancer
* Active TB

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Schiff, MD, Study Director
Locations (12):
- United States (12):
  - Rheumatology Associates of N. Alabama, Huntsville, Alabama
  - Sun Valley Arthritis Center, Ltd., Peoria, Arizona
  - Arizona Arthritis and Rhematolgy Research, Phoenix, Arizona
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Westroads Medical Group, Omaha, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Buffalo Rheumatology, Orchard Park, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Rheumatology and Immunotherapy Center, Oak Creek, Wisconsin

REFERENCES:
- [Result] Schiff MH, von Kempis J, Goldblum R, Tesser JR, Mueller RB. Rheumatoid arthritis secondary non-responders to TNF can attain an efficacious and safe response by switching to certolizumab pegol: a phase IV, randomised, multicentre, double-blind, 12-week study, followed by a 12-week open-label phase. Ann Rheum Dis. 2014 Dec;73(12):2174-7. doi: 10.1136/annrheumdis-2014-205325. Epub 2014 Jun 27. PMID 24972708
- See also: EULAR 2012 SAT0144 — http://www.EULAR.org
- See also: Schiff,m — http://www.rheumatology.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients recruited from US medical/Rheumatology clinics
Pre-assignment Details: patients excluded from protocol if they did not meet entry criteria for active Rheumatoid arthritis
Groups:
- Active Treatment With Cimzia: Reporting group: Cimzia : prefilled 200mg Cimzia syringes. Cimzia 400mg SC at baseline, weeks 2 and 4 and Cimzia 200mg SC at weeks 6, 8, and 10 during the Double Blind Portion.
  Cimzia 400mg SC at weeks 12, 14, and 16 and Cimzia 200mg SC at weeks 18, 20, and 22.
  27 patients entered the Double Blind Portion.
- Placebo: Reporting group: Placebo : prefilled saline syringe during the Double Blind Period
  10 patients entered
Period: Double Blind Period
Arm/Group | Active Treatment With Cimzia | Placebo
Started | 27 | 10
Completed | 26 | 8
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Open Label Period
Arm/Group | Active Treatment With Cimzia | Placebo
Started | 26 | 8
Completed | 22 | 8
Not Completed | 4 | 0
Not completed — Lack of Efficacy | 3 | 0
Not completed — Subject moved | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment With Cimzia: Cimzia : prefilled 200mg Cimzia syringe SC q 2 weeks
  27 patients entered
- Placebo: Placebo : prefilled saline syringe
  10 patients entered
- Total: Total of all reporting groups
Arm/Group | Active Treatment With Cimzia | Placebo | Total
Number analyzed (Participants) | 27 | 10 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 8 | 31
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 27 | 10 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a Clinical Disease Activity Index (CDAI) Decrease of Greater Than or Equal to 10 Points in the Cimzia Treatment Group Compared to the Placebo Group at Week 12
Description: The Clinical Disease Activity (CDAI)is a composite score. Clinical Disease Activity (CDAI) = SJC(28): Swollen 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs (including thumb IP)+ TJC(28): Tender 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs (including thumb IP)+ PGA: Patient Global disease Activity (patient's self assessment of overall RA disease activity on a scale 0-10 where 10 is maximal activity)+ EGA: Evaluator's Global disease Activity (evaluator's assessment of overall RA disease activity on a scale 0-10 where 10 is maximal activity) Remission: CDAI ≤ 2.8; Low Disease Activity: CDAI > 2.8 and ≤ 10 ;Moderate Disease Activity: CDAI > 10 and ≤ 22; High Disease Activity: CDAI > 22. A CDAI reduction of 6.5 represents moderate improvement.
Time Frame: Baseline to week 12
Population: 35 subjects were included in the efficacy assessment at week 12. Subjects in the efficacy assessment at week 12 completed at least 4 weeks of dosing
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 26 | 9
participants | 22 | 2

2. Secondary Outcome: Proportion of Subjects Achieving an American College of Rheumatology 50% (ACR50) Response Criteria in the Cimzia Treatment Group Compared to the Placebo Group at Week 12
Description: ACR50 responders are subjects with at least 50% improvement from baseline for tender joint cout (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale.
  HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do.
  Visual Analog Scale (VAS) - assessment of arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 26 | 9
participants | 5 | 0

3. Secondary Outcome: Proportion of Subjects Achieving an American College of Rheuamtology Low Disease Activity Score and/or Remission Score in the Cimzia Group Compared to the Placebo Group as Calculated by DAS28 (CRP)
Description: The Disease Activity Score-28-C-reactive Protein (DAS28-CRP)is a composite measure for rheumatoid arthritis (RA) is based on 4 variables: tender and swollen joint counts (28 joints),C-Reactive Protein(CRP), and patient global assessment visual analog scale. A lower score indicated less disease activity.
  Remission: CDAI ≤ 2.8; Low Disease Activity: CDAI > 2.8 and ≤ 10 ;Moderate Disease Activity: CDAI > 10 and ≤ 22; High Disease Activity: CDAI > 22
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 26 | 9
participants | 6 | 0

4. Primary Outcome: Proportion of Subjects Achieving an American College of Rheumatology 20% (ACR20) Response Criteria in the Cimzia Treatment Group Compared to the Placebo Group
Description: ACR20 responders are subjects with at least 20% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale(VAS).
  HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do.
  Visual Analog Scale (VAS) - assessment of arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: From Baseline to Week 12
Population: 35 subjects were included in the efficacy assessment at week 12. Subjects in the efficacy assessment at week 12 completed at least 4 weeks of dosing. 30 subjects who completed the 24 week study were included in the efficacy assessment at week 24.
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 26 | 9
participants | 16 | 0

5. Secondary Outcome: Proportion of Subjects Achieving a EULAR Good or Moderate Response Criteria in the Cimzia Treatment Group Compared to the Placebo Group
Description: The EULAR (European League Against Rheumatism) response criteria is a classified response criteria which classifies the patients individual as non-, moderate or good responders dependent on the change and the level of the Disease Activity Score.
  The Disease Activity Score(DAS28) is a continuous disease measure composite of 4 variables: 28 tender joint count, 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. High disease activity= > 5.1, low disease activity= < 3.2, and remission= < 2.6. Clinically significant response= decrease of >1.2 from baseline. Utilizing EULAR response criteria, DAS28 categorical responses define a good (absolute: <3.2 or >1.2 improvement from baseline), moderate (absolute: 3.2-5.1 or 0.6-1.2 change from baseline), or no response (absolute: >5.1 or <0.6 change from baseline).
Time Frame: Baseline to week 12
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 26 | 9
participants | 17 | 0

6. Secondary Outcome: Proportion of Subjects Achieving a CDAI Score Decrease Greater Than or Equal to 13.9 Points in the CimZia Treatment Group Compared to the Placebo Group at Week 12
Description: as for outcome 1
Time Frame: Baseline to week 12
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 26 | 9
participants | 17 | 0

7. Other Pre Specified Outcome: Proportion of Subjects Achieving a CDAI Decrease of Greater Than or Equal to 10 Points in the Cimzia Treatment Group Compared to the Placebo Group at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: 30 subjects were included in the efficacy assessment as week 24. Subjects completed 24 weeks dosing including a 12 week open-label phase.
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 22 | 8
participants | 18 | 6

8. Other Pre Specified Outcome: Proportion of Subjects Achieving an American College of Rheumatology 20% (ACR20) Response Criteria in the Cimzia Treatment Group Compared to the Placebo Group
Description: ACR20 responders are subjects with at least 20% improvement from baseline for tender joint cout (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale.
  HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do.
  Visual Analog Scale (VAS) - assessment of arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline to Week 24
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 22 | 8
participants | 12 | 5

9. Other Pre Specified Outcome: Proportion of Subjects Achieving an American College of Rheumatology 50% (ACR50) Response Criteria in the Cimzia Treatment Group Compared to the Placebo Group
Description: as for outcome 2
Time Frame: Baseline to Week 24
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 22 | 8
participants | 6 | 3

10. Other Pre Specified Outcome: Proportion of Subjects Achieving an American College of Rheuamtology Low Disease Activity Score and/or Remission Score in the Cimzia Group Compared to the Placebo Group as Calculated by DAS28 (CRP)
Description: as for outcome 3
Time Frame: Baseline to Week 24
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 22 | 8
participants | 7 | 3

11. Other Pre Specified Outcome: Proportion of Subjects Achieving a EULAR Good or Moderate Response Criteria in the Cimzia Treatment Group Compared to the Placebo Group
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 22 | 8
participants | 17 | 6

12. Other Pre Specified Outcome: Proportion of Subjects Achieving a CDAI Score Decrease Greater Than or Equal to 13.9 Points in the CimZia Treatment Group Compared to the Placebo Group at Week 24
Description: The Clinical Disease Activity (CDAI)is a composite score. Clinical Disease Activity (CDAI) = SJC(28): Swollen 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs (including thumb IP)+ TJC(28): Tender 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs (including thumb IP)+ PGA: Patient Global disease Activity (patient's self assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity)+ EGA: Evaluator's Global disease Activity (evaluator's assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity) Remission: CDAI ≤ 2.8; Low Disease Activity: CDAI > 2.8 and ≤ 10 ;Moderate Disease Activity: CDAI > 10 and ≤ 22; High Disease Activity: CDAI > 22. A CDAI reduction of 6.5 represents moderate improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Active Treatment With Cimzia | Placebo
Number analyzed (Participants) | 22 | 8
participants | 16 | 5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time informed consent was signed through the whole study period of 24 weeks. In addition, serious adverse events were collected up to 4 weeks after completion/discontinuation of the study.
Description: As refer to the Safety Set which included all subjects who received at least 1 dose of study medication. Active treatment with Cimzia included those subjects in the double-blind portion of the protocol as well as the open label portion of the protocol.
Arm/Group | Active Treatment With Cimzia | Placebo
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/10
Other Adverse Events (participants affected / at risk) | 27/34 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment With Cimzia (N=34) | Placebo (N=10)
gastric ulcer bleed (Gastrointestinal disorders) | 1 | 0 — Subject hospitalized after the last visit of the protocol but prior to the 30 day follow-up phone call.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Active Treatment With Cimzia (N=34) | Placebo (N=10)
upper respiratory infections (Infections and infestations) | 5/27 (5) | 0 (0)
cough (Infections and infestations) | 3 (3) | 1 (1)
tooth abcess (Infections and infestations) | 1 (1) | 0 (0)
cold sore (Infections and infestations) | 2 (2) | 0 (0)
head congestion (General disorders) | 1 (1) | 1 (1)
sinus infection (Infections and infestations) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
fever (Infections and infestations) | 1 (1) | 0 (0)
spider bite (Infections and infestations) | 1 (1) | 0 (0)
sore throat (Infections and infestations) | 1 (1) | 1 (1)
bronchitis (Infections and infestations) | 3 (3) | 0 (0)
viral cold (Infections and infestations) | 2 (2) | 0 (0)
athletes foot (Infections and infestations) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0)
mouth sores (Infections and infestations) | 1 (1) | 0 (0)
third degree burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
actenic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
oral thrush (Infections and infestations) | 1 (1) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 1 (1)
hot face (General disorders) | 1 (1) | 0 (0)
increased knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
back strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
shingles (Infections and infestations) | 1 (1) | 0 (0)
heel pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
gastrointestinal virus (Gastrointestinal disorders) | 2 (2) | 0 (0)
allergies (General disorders) | 1 (1) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
sinus congestion (Infections and infestations) | 1 (1) | 0 (0)
rhinorrhea (Infections and infestations) | 1 (1) | 0 (0)
conjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
shoulder sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle tenderness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
coronary disease (Cardiac disorders) | 1 (1) | 0 (0)
kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
hand pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
bruised tailbone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
fall (General disorders) | 1 (1) | 0 (0)
swollen elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
rheumatoid arthritis flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
chest congestion (Infections and infestations) | 1 (1) | 0 (0)
bug bites (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less